CLINICAL TRIAL: NCT06549894
Title: Evaluation of Biomechanical Forced During the Practice of Endoscopic Submucosal Dissection
Acronym: ENDERGO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Hospices Civils de Lyon (Other); University Hospital, Lille (Other); Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PI2024_843_0031
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Endoscopic Submucosal Dissection; Physiology; Musculoskeletal Disorders
Keywords: Endoscopic submucosal dissection; biomechanic; physiology; Musculoskeletal Disorders
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Performing endoscopic examinations — Performing endoscopic examinations in the conventional framework of patient follow-up. No patient data is collected. The physician performing the act is the subject of the study.

SUMMARY:
The prevalence of musculoskeletal disorders (MSDs) among endoscopists is estimated between 29 and 89%. The most common disorders are carpal tunnel syndrome, De Quervain tenosynovitis, lateral epicondylitis and neck pain. Factors associated with MSD among gastroenterologists practicing endoscopy are: the high number of procedures (more than 20/week), the procedure time (more than 16 hours/week) and the number of years of practice.With the evolution of digestive endoscopy superficial cancer can endoscopically be removed by endoscopic submucosal dissection (ESD) avoiding surgical resections. The number of procedures is increasing, with longer examination times in case of ESD (about 2 hours). This volume of hours and procedures may in the near future further increase the risk of MSDs in the population of gastroenterologists. Some good practice recommendations have been proposed to improve practitioner comfort, similar to what is recommended for digestive surgeons. It is recommended to use a height-adjustable examination table, position the screen at eye level, and use a seat during the procedure. There is little data on the biomechanical forced experienced by an endoscopist when performing endoscopy and colonoscopy, and none when performing ESD.

The aim of this study is to evaluate the biomechanical forced experienced by the gastroenterologist during an ESD the practice of submucosal dissection.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject (age ≥ 18 years)
* hepato-gastroenterologist
* hepato-gastroenterologist performing endoscopic submucosal dissection
* Person who has given consent for participation in the study

Exclusion Criteria:

* non hepato-gastroenterologist
* Person who has not given consent for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
variation of muscle angular during submucosal dissection | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire d'Amiens, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No